CLINICAL TRIAL: NCT06220422
Title: Assessment the Benefit of a Service Procedure Management of NACO in the Treatment of Fractures of the Upper Extremity of the Femur
Brief Title: Assessment of a Procedure for Managing Oral Anticoagulants (NACO) in the Management of Fractures
Acronym: STOP-NACO
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD0123
Record Dates: First submitted 2024-01-03; First posted 2024-01-24 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Femur Fracture
Keywords: NACO; Fracture; Upper end of the femur; Department new procedure
MeSH Terms: conditions — Femoral Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard Department procedure for managing direct-acting oral anticoagulants: Standard Department procedure for managing direct-acting oral anticoagulants (NACO < 50 ng/mL) in the management of fractures before September 2021
  Interventions: Procedure: Standard Department procedure for managing direct-acting oral anticoagulants
- New Department procedure for managing direct-acting oral anticoagulants: Intervention Description New Department procedure for managing direct-acting oral anticoagulants (NACO < 100 ng/mL) in the management of fractures after September 2021
  Interventions: Procedure: New Department procedure for managing direct-acting oral anticoagulants

INTERVENTIONS:
Procedure: Standard Department procedure for managing direct-acting oral anticoagulants — Standard Department procedure for managing direct-acting oral anticoagulants (NACO < 50 ng/mL) in the management of fractures before September 2021
  Groups: Standard Department procedure for managing direct-acting oral anticoagulants
Procedure: New Department procedure for managing direct-acting oral anticoagulants — New Department procedure for managing direct-acting oral anticoagulants (NACO < 100 ng/mL) in the management of fractures after September 2021
  Groups: New Department procedure for managing direct-acting oral anticoagulants

SUMMARY:
The purpose of this study is to demonstrate that by allowing patients with an anticoagulant level less than 100 ng/ml to have their fracture managed surgically, will reduce the delay in surgery and therefore the complications associated. It will also demonstrate that there are no more complications with this new management than from remaining with a bleeding fracture.

DETAILED DESCRIPTION:
Fracture of the upper extremity of the femur are constantly on the increase and represent a public health issue in a population with increasing life expectancy. In the majority of cases, this fracture requires rapid surgical treatment, ideally within 48 hours, before complications, associated with the supine position, appear. A prolonged surgical delay is responsible for multiple complications and increase mortality in a potentially comorbid and fragile population.

Oral anticoagulants (NACOs) are now widely used in general population for cardiovascular diseases, such as non-valvular atrial fibrillation or thrombo-embolic events. Their activity and circulation rate are assessed by an Anti-Xa assay. The current recommendation for scheduled surgery is an assay with an anti-Xa activity of less than 50 ng/mL.

The acquisition of this assay and the wait for a decrease in anti-Xa activity are currently a factor of lengthening the surgical delay leading to proposal a new dosage. By offering the possibility of surgical management with an anti-Xa activity of less than 100 ng/ml, the purpose is to demonstrate a reduction in surgical delay (less than 48 hours) and associated complications. One of the secondary purposes is also to demonstrate that there are no more intra and post-operative complications with this new protocol.

ELIGIBILITY:
Inclusion Criteria :

* Patients on NACO undergoing surgery for fracture of the upper end of the femur,
* 18 years and over,
* Informed patients who did not object.

Exclusion Criteria :

* Patients under court protection,
* Patients under guardianship/curators .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on new anticoagulants undergoing surgery for fracture of the upper end of the femur between 2018 and 2023
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Highlighting of a reduction in the time to surgical management of fracture of the upper end of the femur by adjusting the preoperative threshold for the dosage of of direct-acting oral anticoagulants | At the end of the study, an average of 1 month
  Comparison of time from hospital admission to surgery (in hours) between both groups

SECONDARY OUTCOMES:
Measure of the impact of the department's new strategy (NACO threshold < 100 ng/mL) on estimated intraoperative blood loss | At the end of the study, an average of 1 month
  Comparison on the amount of blood lost (mL) between both groups
Description of the impact of the department's new strategy (NACO threshold < 100 ng/mL) on transfusion requirement | At the end of the study, an average of 1 month
  The impact on transfusion requirements between both groups is evaluate on the following items :
  * Packed red blood cells,
  * Fresh frozen plasma,
  * Unit concentrate of platelets,
  * 4-factor prothrombin complex concentrate.
Description of the impact of the department's new strategy (NACO threshold < 100 ng/mL) on the hospital morbidity | At the end of the study, an average of 1 month
  The impact on Hospital morbidity between both groups is evaluate on the following complications :
  * Infectious complications (surgical site infection, nosocomial infections: urinary, pneumonia, others),
  * Thromboembolic complications (pulmonary embolism, deep vein thrombosis),
  * Cardiovascular complications (decompensation of heart failure, Acute pulmonary oedema, ACS),
  * Post-operative haemorrhagic complications (surgical site haematoma requiring treatment),
  * 30-day readmission
Measure the impact of the department's new strategy (NACO threshold < 100 ng/mL) on the hospital mortality | At the end of the study, an average of 1 month
  Comparison on the number of deaths in each group.
Measure of the impact of the department's new strategy (NACO threshold < 100 ng/mL) on the complications affecting surgical management | At the end of the study, an average of 1 month
  The impact on the factors affecting surgical management between both groups is evaluate on the following item :
  - Complications of the supine position (bedsores, etc.) and those related to the field (confusion, physical restraint indwelling catheter, stay in intensive care, resumption walking /chair, delay in returning home, Follow-up care and rehabilitation (SSR), geriatric assessment, nutritional management)
Measure of the impact of the department's new strategy (NACO threshold < 100 ng/mL) on the degree of dependence due to surgical management | At the end of the study, an average of 1 month
  The impact on the factors affecting surgical management between both groups is evaluate on the following item :
  - Degree of dependence according to the Katz evaluation scale, The KATZ scale is used to determine the degree of dependency of patients. It consists of a questionnaire assessing their abilities in 6 areas of daily life. For each area, the response varies between 4 scores ranging from no assistance to the need for total assistance.
Measure of the impact of the department's new strategy (NACO threshold < 100 ng/mL) on the factors affecting surgical management | At the end of the study, an average of 1 month
  The impact on the factors affecting surgical management between both groups is evaluate on the following item :
  - Day of admission to care (weekend/holiday/on-call day)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Amélie TOUSSAINT, Principal Investigator — Hôpital NOVO
Locations (1):
- Anaesthetics department - Hôpital NOVO - Pontoise Site, Pontoise, France